CLINICAL TRIAL: NCT01654120
Title: Liraglutide and Insulin-001 A Randomized Prospective Trial of Liraglutide Added to High-Dose Insulin Therapy vs. High-Dose Insulin Therapy Alone in Insulin-Resistant Patients With Type 2 Diabetes
Brief Title: Study of Effectiveness of Liraglutide Added to High Dose Insulin in Type II Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mountain Diabetes and Endocrine Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: high dose and lira 001
Record Dates: First submitted 2011-12-16; First posted 2012-07-31 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type II
Keywords: insulin; Type II Diabetes; liraglutide; Glucagon-Like Peptide 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Liraglutide; Insulin; Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide plus insulin (Experimental): Patients were randomized to receive liraglutide plus insulin (LIRA) for 12 months.
  Interventions: Drug: Liraglutide; Drug: Insulin
- Insulin titration only (Active Comparator): Patients were randomized to receive insulin only (control) for 6 months. The controls were then crossed over to receive liraglutide plus insulin for 6 months after the initial control period.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Liraglutide — SC, 1.8mg,QD, six months to one year
  Other Names: Victoza
  Arms: liraglutide plus insulin
Drug: Insulin — SC, will be titrated during the study, 4 times a day, 1 year
  Other Names: U-500; Levemir; Novolog

SUMMARY:
The purpose of this study is to determine the effect of adding liraglutide to high dose insulin therapy compared to high dose insulin therapy alone in patients with insulin-treated Type 2 diabetes with insulin requirements of > 100 units of insulin per day.

DETAILED DESCRIPTION:
40 subjects with Type 2 diabetes using > 100 units of insulin per day with or without metformin with HbA1c > 6.5% will be randomized into 2 treatment groups: treatment group will have liraglutide added to insulin and control group will have insulin uptitration only for 6 months. Primary endpoint to be compared between groups will be HbA1c at 6 months. Secondary endpoints will include weight, total daily insulin dose, percent time in euglycemic, hyperglycemic, and hypoglycemic ranges by continuous glucose monitor (CGM), and effect on GlycoMark and hs-CRP. Safety endpoints will include incidence of hypoglycemia and incidence of gastrointestinal side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with Type 2 diabetes with HbA1c from 6.5 to 10% treated with intensive insulin therapy (MDI or CSII, including U-500 insulin-treated patients) using > 100 units of insulin, with or without a stable dose of oral insulin sensitizing medications, for at least three months.
2. Aged 18 to 80 years.
3. Females of child-bearing potential must be using adequate form of contraception.
4. Patient willing to monitor BG four times daily, use CGM, and comply with study-related protocol.

Exclusion Criteria:

1. Type 1 diabetes.
2. Use of any GLP-1 receptor agonist within previous three months.
3. Use of DPP-4 inhibitors or oral insulin secretagogues within the previous three months.
4. Use of glucocorticoids (except inhaled).
5. Use of any experimental drug within previous three months.
6. Known or suspected allergy to liraglutide, Novolog or Levemir.
7. Personal or family history of medullary carcinoma of the thyroid or MEN-2.
8. Concomitant chronic renal disease with creatinine > 1.5%.
9. Concomitant chronic hepatic, gastrointestinal or other illness (including pancreatitis or active cardiovascular disease except stable exertional angina).
10. Inability or unwillingness to monitor BG, use CGM, or comply with study protocol.
11. Women of child-bearing potential unwilling to use adequate contraception, intending to become pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at six months | baseline and six months
  Glycemic control as measured by HbA1c

SECONDARY OUTCOMES:
Hypoglycemia | 6 months and 12 months
  The frequency and severity of hypoglycemia in each treatment arm by glucose meter download and by percent time spent in the hypoglycemic range (BG < 70 mg/dl) by CGM will be assessed at six and 12 months
Total Daily Insulin Dose (TDID) | 3, 6, 9, and 12 months
  TDID will be determined in each treatment arm for statistical comparisons at three and six months, and for entire cohort at nine and 12 months.
Weight | baseline, 3, 6, 9, and 12 months
  Weight will be statistically compared to baseline and between treatment arms at three and six months, and for entire cohort between baseline, six, nine and 12 months.
GlycoMark | baseline, 3, 6, 9, and 12 months
  Postprandial glycemic control as assessed by GlycoMark and CGM will be compared between study groups at three and six months, and for entire cohort compared to baseline at nine and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy S Lane, MD, Principal Investigator — Mountain Diabetes and Endocrine Center
Locations (1):
- Mountain Diabetes and Endocrine Center, Asheville, North Carolina, United States